CLINICAL TRIAL: NCT06612710
Title: An Open-label Exploratory Clinical Trial to Assess the Safety and Efficacy of NouvSoma001 in the Treatment of Ischemic Stroke
Brief Title: The Safety and Efficacy of NouvSoma001 in Ischemic Stroke
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wei Wang (Other)
Collaborators: iRegene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Wei Wang, Prof., Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NouvSoma001inIS
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; extracellular vesicles
MeSH Terms: conditions — Ischemic Stroke | interventions — Injections, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extracellular vesicles group (Experimental): Patients in this arm will be given extracellular vesicles derived from human-induced neural stem cells for intravenous injection once a day for 7 days.
  Interventions: Drug: extracellular vesicles derived from human induced neural stem cell for intravenous injection
- extracellular vesicles placebo group (Placebo Comparator): Patients in this arm will be given a placebo of extracellular vesicles derived from human-induced neural stem cells for intravenous injection once a day for 7 days.
  Interventions: Drug: a placebo of extracellular vesicles derived from human induced neural stem cell for intravenous injection

INTERVENTIONS:
Drug: extracellular vesicles derived from human induced neural stem cell for intravenous injection — extracellular vesicles derived from human induced neural stem cell for intravenous injection（4×10^9 particles/kg）
  Other Names: NouvSoma001
  Arms: extracellular vesicles group
Drug: a placebo of extracellular vesicles derived from human induced neural stem cell for intravenous injection — extracellular vesicles placebo (4×10^9 particles/kg)
  Other Names: NouvSoma001placebo
  Arms: extracellular vesicles placebo group

SUMMARY:
This is a single-center, randomized, open-label, placebo-controlled, dose-escalation trial. The objective of this research is to evaluate the safety, tolerability, and preliminary efficacy of intravenous administration of human-induced neural stem cell-derived extracellular vesicles (NouvSoma001) in the treatment of ischemic stroke.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, placebo-controlled, dose-escalation trial. This study will consist of 2 parts, with Part 1 being a dose-escalation study and Part 2 being a dose-extension study based on the results of Part 1. Part 1 will follow a traditional 3+3 dose-escalation design, enrolling a total of 9 subjects. Cohort 1: receive 4×10^9 particles/kg, Cohort 2: receive 8×10^9 particles/kg, and Cohort 3: receive 1.6×10^10 particles/kg. If no dose-limiting toxicities (DLT) are observed within 2 weeks after the initial administration, a new cohort will be enrolled at the next higher dose level. If DLTs are observed in 1 participant, another 2 participants will be treated at the same dose level. Dose escalation will cease if DLTs are observed in more than 33% of the participants. In Part 2, the remaining 60 participants will be randomized in a 2:1 ratio to the treatment and placebo groups, with the dose level determined by the Data Safety Monitoring Board based on the results of Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the recruiters ranged from 18 to 75 years.
2. Clinical diagnosis of ischemic stroke, the time of stroke onset is known, and the onset occurred no more than 7 days before enrollment.
3. Magnetic resonance imaging (MRI) or computed tomography (CT) findings consistent with ischemic stroke.
4. At the time of enrollment, the NIHSS score is between 6 and 20; additionally, there is at least one limb with muscle strength ≤ Grade 3.
5. Patients who have the mental capacity to understand and participate in the study.
6. Informed consent was obtained from patients or their legal representatives.

Exclusion Criteria:

1. CT indicates intracranial hemorrhage, including hemorrhagic stroke, epidural hematoma, subdural hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, or hemorrhagic transformation.
2. Patients with Alzheimer's disease, Parkinson's syndrome, or other neurodegenerative disorders.
3. Evidence of brain tumors, epilepsy, or a history of traumatic brain injury.
4. Presence of non-vascular diseases causing white matter lesions, such as carbon monoxide poisoning, multiple sclerosis, or adrenoleukodystrophy.
5. Rapid spontaneous neurological improvement during the screening period, defined as a reduction of NIHSS score by ≥ 8 points from symptom onset to the first administration.
6. Persistent systemic infection, severe local infection, or ongoing use of immunosuppressants.
7. Patients with malignant diseases or an expected survival of less than 5 years.
8. Significant hearing or vision impairments, language disorders, or claustrophobia that would hinder cooperation with neuropsychological assessments and MRI examinations.
9. Contraindications to MRI.
10. Patients unable to comply with follow-up requirements during the study.
11. Severe liver, renal, cardiac, or pulmonary insufficiency, hematologic disorders, or malignant tumors (Liver insufficiency is defined as ALT or AST levels greater than 1.5 times the upper normal limit; renal insufficiency is defined as serum creatinine levels greater than 1.5 times the upper normal limit).
12. Patients with alcohol addiction or those testing positive for drug abuse.
13. Patients with a history of severe allergies or known allergy to human biological products.
14. Pregnant or breastfeeding women, and those planning to conceive during the trial period.
15. Participation in other clinical trials within the past 3 months.
16. Patients considered unsuitable for participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of all adverse events (AE) and serious adverse events (SAE) | Up to 6 month after treatment initiation
  The assessment of adverse events and serious adverse events

SECONDARY OUTCOMES:
The incidence and severity of all adverse events (AE) and serious adverse events (SAE) | Up to 18 month after treatment initiation
  The assessment of adverse events and serious adverse events
Magnetic Resonance Imaging(MRI) at month 3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The National Institutes of Health Stroke Scale, NIHSS | Up to 6 month after treatment initiation
  To assess NIHSS of subjects at month 1、3、6 after treatment initiation
The Modified Rankin Scale (mRS) | Up to 6 month after treatment initiation
  To assess mRS of subjects within month 1、3、6 after treatment initiation
The score of Mini-mental State Examination (MMSE) at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of MMSE ranges from 0 to 30, and 30 represents the best.
The score of Montreal cognitive assessment scale (MoCA) at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of MoCA ranges from 0 to 30, and 30 represents the best.
The score of Barthel Index for activities of daily living (ADL) at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of ADL ranges from 0 to 100, and 100 represents the best.
The score of Hamilton Depression Scale at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of Hamilton Depression Scale ranges from 0 to 81, and 81 represents the worst.
The score of Hamilton Anxiety Scale at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of Hamilton Anxiety Scale ranges from 0 to 56, and 56 represents the worst.
The score of Clock Drawing Test at month 1、3、6 compared with baseline and control group | Up to 6 month after treatment initiation
The value of Quality of Life (EQ-5D-5L) at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The score of Alzheimer's disease assessment scale-cognitive section (ADAS-cog) at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of Alzheimer's disease assessment scale-cognitive section ranges from 0 to 70, and 70 represents the worst.
The score of Clinical Dementia Rating (CDR) at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The score of Hopkins verbal learning test（HVLT）at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The incidence of Columbia-Suicide Severity Rating Scale (C-SSRS) events at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The value of Nfl and GFAP in serum at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, MD, Principal Investigator — Tongji Hospital; Daishi Tian, MD, Principal Investigator — Tongji Hospital; Chuan Qin, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University ofScience and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang R, Mao W, Niu L, Bao W, Wang Y, Wang Y, Zhu Y, Yang Z, Chen J, Dong J, Cai M, Yuan Z, Song H, Li G, Zhang M, Xiong N, Wei J, Dong Z. NSC-derived exosomes enhance therapeutic effects of NSC transplantation on cerebral ischemia in mice. Elife. 2023 Apr 27;12:e84493. doi: 10.7554/eLife.84493. PMID 37104115
- [Result] Zhu ZH, Jia F, Ahmed W, Zhang GL, Wang H, Lin CQ, Chen WH, Chen LK. Neural stem cell-derived exosome as a nano-sized carrier for BDNF delivery to a rat model of ischemic stroke. Neural Regen Res. 2023 Feb;18(2):404-409. doi: 10.4103/1673-5374.346466. PMID 35900437
- [Result] Gao G, Li C, Ma Y, Liang Z, Li Y, Li X, Fu S, Wang Y, Xia X, Zheng JC. Neural stem cell-derived extracellular vesicles mitigate Alzheimer's disease-like phenotypes in a preclinical mouse model. Signal Transduct Target Ther. 2023 Jun 14;8(1):228. doi: 10.1038/s41392-023-01436-1. No abstract available. PMID 37311758